CLINICAL TRIAL: NCT06661603
Title: Effect of Practicing Yoga and Meditation on Cortisol Hormone, Immunoglobulin a and Metabolic Parameter Among Medical Students
Acronym: GSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GSY (Goodbye Stress with Yoga)
Record Dates: First submitted 2024-06-23; First posted 2024-10-28 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Adult Children
Keywords: Medical students; Yoga; Cortisol Hormone; Immunoglobulin; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GSY Yoga Intervention (Experimental): GSY Goodbye Stress with Yoga Protocol Full body warm-up and light stretching exercise 15 min Performing various yoga postures - including standing, sitting, prone, and supine yoga postures (Asanas) 50 min Breathing exercises = (Pranayama)10 min and Meditation15 min
  *The development of the yoga protocol, named "GSY Goodbye Stress with Yoga Protocol," was a collaborative effort involving a certified yoga trainer, a medical researcher, and experienced yogis from India.
  Interventions: Behavioral: GSY Yoga Intervention
- Control Group (No Intervention): The participants who don't receive any kind of therapy, which means the control group with standard care and without any treatment or intervention.

INTERVENTIONS:
Behavioral: GSY Yoga Intervention — In the GSY yoga intervention, where participants received 90 minutes/week yoga intervention for duration of 10 weeks.
  Arms: GSY Yoga Intervention

SUMMARY:
This clinical trial aims to develop and test a yoga intervention to improve cortisol hormone rhythm, immunoglobulin A, and metabolic markers among medical students. The development of the yoga protocol, "GSY Goodbye Stress with Yoga Proto-col," was a collaborative effort involving a certified yoga trainer, medical researcher, and experienced yogis from India. GSY yoga intervention, which includes yoga asanas poses, breathing techniques, and guided meditation, may reduce stress levels, improve immunity, and enhance other metabolic parameters in medical students.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1. To examine the effectiveness of yoga intervention as a stress reduction technique and measure its effects on the level of cortisol, immunoglobulin A (IgA), and metabolic parameters.
2. To Compare the outcomes of a yoga intervention group to a non-yoga intervention group to determine whether practicing yoga can reduce the negative impacts of elevated cortisol on the physiological parameters.

SECONDARY OBJECTIVES:

1. To determine the correlation between the psychophysiological stress and cortisol hormone in students.
2. To investigate the effect of yoga intervention on student mental health and well-being.

OUTLINE:

Participants receive yoga intervention from a certified yoga trainer once a week for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the study required participants to be currently enrolled in the Medicine Faculty of the University of Pecs

Exclusion Criteria:

Students with illnesses (such as recent injuries, chronic pain, or significant arthritis) that would make it unsafe for them to take part in a yoga intervention will be excluded from the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Effect of GSY Yoga Intervention in the Improvement of Immunoglobulin A among Medical Students | upto 10 weeks
  Samples of saliva cortisol will be collected to analyse diurnal cortisol rhythm , at the beginning and the end of the first and the last yoga class to determine immediate and longitudinal effects and to measure the diurnal rhythms of immunoglobulin.
Efficacy of GSY yoga intervention in the reduction of cortisol hormone rhythm | upto 10 weeks
  Samples of saliva cortisol will be collected, at the beginning and the end of the first and the last yoga class to determine immediate and longitudinal effects and to measure the diurnal rhythms of cortisol.
Efficacy of GSY yoga intervention in the cortisol hormone by using hair cortisol concentration | 10 weeks
  Samples of hair cortisol will be collected to measure hair cortisol concentration for analyzing the long-term cortisol level in individuals, at the beginning and the end of the first and the last yoga class
Effect of 10 weeks yoga intervention on immune and metabolic parameter among medical students | Upto 10 weeks
  Blood sample will be collected to analyse Immune parameter, including Immunoglobulin A, Immunoglobulin G, Immunoglobulin M, and Metabolic parameter including, Fasting Blood Glucose FBG, HBA1C, LDL,HDL,total cholesterol, triglycerides, and non-HDL at the beginning and the end of the first and the last yoga class to determine immediate and longitudinal effects. .

SECONDARY OUTCOMES:
Changes in Quality of life | upto 10 weeks
  The change in the quality of life before and after yoga intervention is measured by collecting data from participants using the WHOQOL (World Health Organization Quality of Life-Bref) tool. The WHOQOL-Bref, a shorter version of the WHOQOL-100, provides a comprehensive measure of quality of life across four domains: physical health, psychological health, social relationships, and environment. Scores for each domain range from 0 to 100, with higher scores indicating a better quality of life.
Changes in sleep quality | upto 10 weeks
  The change in sleep quality before and after the yoga intervention is measured by collecting data from participants using the Pittsburgh Sleep Quality Index (PSQI). The PSQI scores range from 0 to 21, with higher scores indicating worse sleep quality.
Changes in physical activity | upto 10 weeks
  The change in physical activity level before and after the yoga intervention is measured by collecting data from participants using the Global Physical Activity Questionnaire (GPAQ). This tool presents physical activity as a separate outcome measure. the GPAQ scores range in MET( Metabolic Equivalent of Task)-minutes per week, with higher scores indicating higher levels of physical activity.
Changes in stress reduction | upto 10 weeks
  The change in stress levels before and after the yoga intervention is measured by collecting data from participants using the Depression, Anxiety, and Stress Scales (DASS). The DASS scores range from 0 to 42 for each subscale (Depression, Anxiety, Stress), with higher scores indicating greater severity of symptoms.
Changes in emotional regulation | upto 10 weeks
  The change in emotional regulation before and after yoga intervention is measured by collecting data from participants using the DERS (The Difficulties in Emotion Regulation Scale). DERS is an instrument measuring emotion regulation problems. tool.
Changes in Sedentary Behaviour | Upto 10 weeks
  The changes in the sedentary behavior of the participants before and after the yoga intervention will be analyzed by using the Sedentary Behavior Questionnaire (SBQ).

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Chauhan, Principal Investigator — Assistant Professor, PhD student University of Pécs
Locations (1):
- University of Pécs, Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chauhan S, Babu AM, Galgalo DA, Melczer C, Premusz V, Karsai I. Effect of yoga in medical students to reduce the level of depression, anxiety, and stress: pilot study (Goodbye Stress with Yoga GSY). BMC Complement Med Ther. 2024 May 24;24(1):203. doi: 10.1186/s12906-024-04496-0. PMID 38790041
- [Derived] Chauhan S, Najaf SS, Nagy Z, Al-Jawarneh M, Nagy T, Miseta A, Premusz V, Karsai I. An exploratory study on the changes in immune and metabolic parameters by 10 weeks of yoga intervention among medical students. Sci Rep. 2025 Nov 5;15(1):38730. doi: 10.1038/s41598-025-22421-4. PMID 41193511
- [Derived] Chauhan S, Najaf SS, Gergely L, Kinga KA, Karsai I, Premusz V. Impact of 10 Weeks of Yoga Intervention on Mental Health and Overall Well-Being Among Medical Students: GSY Study. Sports (Basel). 2025 Apr 10;13(4):114. doi: 10.3390/sports13040114. PMID 40278740
- See also: Pilot Study Results — https://pubmed.ncbi.nlm.nih.gov/38790041/